CLINICAL TRIAL: NCT06242743
Title: Effect of Needle Bevel Type on Pain Perception in Children During Inferior Alveolar Nerve Block Anesthesia (a Randomized Controlled Clinical Trial)
Brief Title: Type of Needle Bevel on Pain Perception in Children During Inferior Alveolar Nerve Block Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0726_07/2023
Record Dates: First submitted 2024-01-01; First posted 2024-02-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: Scalpel blade needles
- Control group (Active Comparator)
  Interventions: Other: standard blade needles

INTERVENTIONS:
Other: Scalpel blade needles — Patients were assigned to IANB injection by double scalpel blade bevel needles.
  Arms: Test group
Other: standard blade needles — Patients were assigned to IANB injection by standard blade bevel needles.
  Arms: Control group

SUMMARY:
fear of the discomfort that comes with anesthetic needle insertion. For dental local anesthesia, needles with a scalpel-designed bevel have been claimed to decrease pain elicited by injection.

Objective of the study: The purpose of this study is to assess the effect of needle bevel on patient's perception of pain during inferior alveolar nerve block anesthesia and the needle tip will be further assessed for deformation.

Materials and Methods: The study will be a double-blind randomized controlled clinical trial, with a parallel design. A total of sixty-six healthy children will be selected from The Pediatric Dentistry and Dental Public Health Clinic, Faculty of Dentistry, Alexandria University, Egypt. Children will be selected with scores 3 or 4 Frankel behavioral rating scale. Written consent will be obtained from the legal guardian. Participants will be randomly allocated into two groups according to the type of needle bevel that will be used. Group I (test group) will receive inferior alveolar nerve block (IANB) using a double scalpel blade bevel needle, while group II (control group) will receive IANB using a standard blade bevel needle. All the procedures will be videotaped. Pain reaction will be evaluated subjectively using a face scale modified from the Maunuksela scale and objectively using the Sensory, Eye, and Motor (SEM) scale. After the respective single injection, the needles will be fixed on an object slide and prepared for microscopic examination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with ASA I, II Classification.
* Children with no learning disabilities.
* Positive or definitely positive behavior according to the Frankl Scale.
* Patient requiring local anesthetic injection IANB for dental treatment.
* Written consent of the legal guardian.

Exclusion Criteria:

* Medically compromised patient.
* Children with emergency treatment needs, such as abscess, cellulitis and space infection.
* Hypersensitivity to local anesthetic drugs

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Objective Pain assessment | During procedure
  Sound, Eye, and Motor scales will be used for pain assessment by viewing the recorded videotapes for the patients during the dental procedure.
  it assesses changes in comfort level as follows;
  1. Comfort
  2. Mild discomfort
  3. Moderate discomfort
  4. Severe discomfort higher scores mean higher discomfort Minimum score: 1 Maximum score: 12
Subjective pain assessment | During procedure
  Each patient will be trained on using the scale by modeling and then requesting every patient to think of the last time she/he went through a painful experience and to choose the facial expression that best relates his/her current experience of discomfort to the previous one.
  Facial scales' categories are as follows Score A: Satisfied Score B Indifference Score C: Dissatisfaction

SECONDARY OUTCOMES:
Needle deformation | During procedure
  Needles will be evaluated under stereoscopic microscope to measure the amount of deformation or deviation in micorn meter from the original unused ones.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt